CLINICAL TRIAL: NCT06764849
Title: Minimally Invasive Open Excisional Hemorrhoidectomy Compared to Conventional Open Excisional Hemorrhoidectomy: a Clinical Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It corresponds to IDEAL Framework stage 4 and now we are conducting stage 2
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Ignacio Fernandez Hurtado, GENERAL SURGERY SPECIALIST, Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IB5478/24
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hemorrhoidectomy; Hemorrhoids Third Degree; Hemorrhoidal Disease; Postoperative Pain
Keywords: hemorrhoidal disease; minimally invasive open excisional hemorrhoidectomy; open excisional hemorrhoidectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPEN EXCISIONAL HEMORRHOIDECTOMY (Active Comparator): Patients will undergo conventional open excisional hemorrhoidectomy
  Interventions: Procedure: CONVENTIONAL OPEN EXCISIONAL HEMORRHOIDECTOMY
- MINIMALLY INVASIVE OPEN EXCISIONAL HEMORRHOIDECTOMY (Experimental): Patients will undergo open excisional hemorrhoidectomy using a minimally invasive technique
  Interventions: Procedure: MINIMALLY INVASIVE OPEN EXCISIONAL HEMORRHOIDECTOMY

INTERVENTIONS:
Procedure: CONVENTIONAL OPEN EXCISIONAL HEMORRHOIDECTOMY — Hemorrhoidectomy performed based on the conventional technique described by Milligan-Morgan
  Arms: OPEN EXCISIONAL HEMORRHOIDECTOMY
Procedure: MINIMALLY INVASIVE OPEN EXCISIONAL HEMORRHOIDECTOMY — Hemorrhoidectomy performed based on the tecnique described by Milligan Morgan, using a minimally invasive approach.
  Arms: MINIMALLY INVASIVE OPEN EXCISIONAL HEMORRHOIDECTOMY

SUMMARY:
This study aims to demonstrate that open excisional hemorrhoidectomy (OEH), when performed using a minimally invasive approach, results in less postoperative pain and comparable outcomes to conventional OEH.

DETAILED DESCRIPTION:
At our hospital, the investigators have developed a new approach to hemorrhoid surgery by modifying the traditional open excisional hemorrhoidectomy. This new method incorporates an image-amplifying device and utilizes microsurgery tools. Preliminary results have shown significant improvement in patients' immediate postoperative pain, with efficacy comparable to conventional methods one year after treatment.

We propose conducting a clinical trial to confirm these initial findings. The study will include two gropus: one undergoing conventional open excisional hemorrhoidectomy (OEH) and the other receiving minimally invasive open excisional hemorrhoidectomy (miOEH). Patients will be randomly assigned to one of these two groups.

The primary outcome of interest will be the level of postoperative pain assessed 10 days after surgery. The secondary outcomes will evaluate the effectiveness of the technique one year post-surgery, measured by the Hemorrhoidal Disease Symptom Score(HDSS) and the Short Health Scale in Hemorrhoidal Disease (SHSHD).

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years.
* Hemorrhoids grade III.
* Surgical indication for hemorrhoidal disease.

Exclusion Criteria:

* Acute hemorrhoidal disease.
* Previous hemorrhoidal surgery.
* Concomitant anal fissure.
* Concomitant anal fistulae.
* Concomitant rectal prolapse.
* Concomitant inflamatory bowel disease or anal cancer.
* Language impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measured with the visual analogic scale | 10 days
  Postoperative pain presented 10 days after the surgical procedure was measured using the visual analogic scale (VAS). Operationally, a VAS is a horizontal line 100 mm long anchored by word descriptors at each end; on the left-hand end, it says "no pain," and on the right-hand end of the line, it says "very severalPostoperative pain was assessed 10 days after the surgical procedure using the visual analog scale (VAS). The VAS consists of a 100 mm horizontal line, with descriptors at each end. The left end is labeled "no pain," while the right end is labeled "very severe pain." Patients indicate their perception of pain by marking a point on the line. The VAS score is then calculated by measuring the distance in millimeters from the left end of the line to pain". The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring millimetres from the left-hand end of the line to the point the patient marks.
Postoperative pain measured by the number of rescue painkillers needed | 10 days
  Postoperative pain presented 10 days after the surgical procedure was measured with the number of rescue painkillers needed during this period. Patients will take the following analgesic regimen: Paracetamol 1 gram every 8 hours and Dexketoprofen 12.5 milligrams every 8 hours alternately. Tramadol 50 milligrams will be used as rescue analgesia. The patient will write down the number of Tramadol tablets needed during the first 10 days on a collection sheetPostoperative pain will be assessed 10 days after the surgical procedure by recording the number of rescue painkillers used during this time. Patients will follow this analgesic regimen: they will take Paracetamol 1 gram every 8 hours and Dexketoprofen 12.5 milligrams every 8 hours, alternating between the two. Tramadol 50 milligrams will be available as rescue analgesia. Patients should note the number of Tramadol tablets taken during the first 10 days on a collection sheet..

SECONDARY OUTCOMES:
Efficacy of the treatment using the Hemorrhoidal Disease Symptom Score | 1 year
  We analyse the efficacy of both procedures using the difference in scores between before and 1 year after surgery on the Hemorrhoidal Disease Symptom Score (HDSS). The HDSS was assessed using the patient-reported frequency of the five symptoms, including pain, itching, bleeding, soiling, and prolapse. Patients were instructed to answer based on their experience during the previous 3 months. Each symptom was graded on a 5-point scale (0 = never, 1 = less than once a month, 2 = less than once a week, 3 = 1-6 days per week, 4 = every day or always), giving a total score ranging from 0 to 20
Efficacy of treatment using the Short Health Scale adapted for hemorrhoidal disease | 1 year
  We analyze the effectiveness of both procedures by comparing the scores on the Short Health Scale adapted for hemorrhoidal disease (SHD-HD) before surgery and one year post-surgery. Patients were asked to report their overall symptom burden, how hemorrhoidal disease interfered with their daily activities, and the concerns it caused them. The fourth question focused on their general well-being. This assessment used a 7-point Likert scale, resulting in a total score that ranges from 4 to 28, with higher values indicating worse health out

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751